CLINICAL TRIAL: NCT07129798
Title: Efficacy and Safety of Myopic Macular Hole Closure Surgery Without Endotamponade Agent
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon KH Szeto, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC/KE-23-0115/ER-4
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Macular Hole; Myopia
Keywords: Macular hole; High Myopia; Vitrectomy; Internal limiting membrane flap; No endotamponade
MeSH Terms: conditions — Retinal Perforations; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ILM flap with no endotamponade technique (Experimental): Patients with myopic macular hole (MH) will undergo pars plana vitrectomy (PPV) and the internal limiting membrane (ILM) flap with no gas tamponade technique to repair the MH.
  Interventions: Procedure: ILM flap with no endotamponade technique

INTERVENTIONS:
Procedure: ILM flap with no endotamponade technique — Standard 3-port pars plana vitrectomy will be performed under either local anesthesia or general anesthesia. After core vitrectomy, posterior vitreous detachment induction will be done using vitrectomy cutter suction with the staining of intravitreal triamcinolone if necessary. This is followed by staining of the ILM with ILM blue dye. A half-moon shaped temporal ILM flap will be created, bridging the MH, using an end-gripping intraocular forceps. The posterior pole would be filled with perfluorocarbon (PFC) liquid and cohesive viscoelastic will be injected under the PFC to stabilize the ILM flap over the MH. Removal of PFC and search for peripheral retinal breaks will be done before removal of vitrectomy trocars and closure of sclerotomies wounds. Surgery will be combined with cataract removal (phacoemulsification) with intraocular lens implantation if patients have visually significant cataract. No specific post-operative posture will be required.

SUMMARY:
Macular hole (MH) is a common condition that affects approximately 1.6/1000 elderly Chinese population. The prevalence is expected to be even higher in individuals with high myopia (HM), an established risk factor for MH. Without prompt surgical intervention, it can lead to irreversible vision loss and retinal detachment. Standard MH surgery involves pars plana vitrectomy (PPV) with internal limiting membrane (ILM peeling), followed by endotamponade agents to appose the MH edge.

Office of Research and Knowledge Transfer Services

Common endotamponade agents include intraocular long-acting gas and silicone oil. The use of endotamponade has its limitations, for example, impairing vision, the need for strict posturing and avoid air travel in the early postoperative period. Ocular complications, such as uveitis, cataract and glaucoma may arise.

To overcome these shortcomings, a novel technique to close MH without endotamponade agents was proposed by a group from Poland. Using viscoelastics to stabilize ILM flap over the MH, negating the need and limitations of endotamponade agents. However, this case series is limited by its small sample size (12 eyes) and lack of patients with pathological myopia (PH).

PH is prevalent in the Asian population and myopic MH tend to have lower surgical success rate due to antero-posterior traction from posterior staphyloma and long axial length associated with PH. There is currently a gap in evidence whether this novel surgical technique could benefit eyes with myopic MH. The investigators plan to conduct a prospective interventional case series to establish the efficacy and safety of myopic MH closure using this novel surgical technique.

DETAILED DESCRIPTION:
Macular hole (MH) is a common condition that affects approximately 1.6/1000 elderly Chinese population. The prevalence is expected to be even higher in individuals with high myopia (HM), an established risk factor for MH. Without prompt surgical intervention, it can lead to irreversible vision loss and retinal detachment. Standard MH surgery involves pars plana vitrectomy (PPV) with internal limiting membrane (ILM peeling), followed by endotamponade agents to appose the MH edge.

Common endotamponade agents include intraocular long-acting gas and silicone oil. The use of endotamponade has its limitations, for example, impairing vision, the need for strict posturing and avoid air travel in the early postoperative period. Ocular complications, such as uveitis, cataract and glaucoma may arise.

To overcome these shortcomings, a novel technique to close MH without endotamponade agents was proposed by a group from Poland. Using viscoelastics to stabilize ILM flap over the MH, negating the need and limitations of endotamponade agents. However, this case series is limited by its small sample size (12 eyes) and lack of patients with pathological myopia (PH).

PH is prevalent in the Asian population and myopic MH tend to have lower surgical success rate due to antero-posterior traction from posterior staphyloma and long axial length associated with PH. There is currently a gap in evidence whether this novel surgical technique could benefit eyes with myopic MH. The investigators plan to conduct a prospective interventional case series to establish the efficacy and safety of myopic MH closure using this novel surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Patients with full thickness macular hole, defined as full thickness foveal defect on OCT
* Patients with pathological myopia, defined as refractive error of </= -6.0D or axial length >/= 26.0mm with signs of posterior staphyloma, lacquer cracks or chorizo-retinal atrophy

Exclusion Criteria:

* Patients with concomitant retinal detachment
* Prior MH surgery
* Macular conditions other than MH, such as myopic choroidal neovascularization, age related macular degeneration and Diabetic Macular Edema
* Patients who cannot be cooperative with ophthalmic examination or give informed consent to undergo surgery
* Fellow eye already recruited in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Macular hole closure rate | 3 months
  Defined as closure of MH on optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Post-operative best-corrected visual acuity | 12 months
  BCVA
MH closure pattern | 12 months
  Grading of MH closure pattern based on OCT

CONTACTS AND LOCATIONS:
Overall Officials: Simon KH Szeto, MBChB, FRCOphth, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Hong Kong Eye Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Need organizational approval

REFERENCES:
- [Background] Szeto SKH, Yu AHY, Tsang CW, Mohamed S, Chen LJ, Lai TYY. COMPLEX MACULAR HOLE CLOSURE BY TEMPORAL INTERNAL LIMITING MEMBRANE FLAP WITHOUT ENDOTAMPONADE. Retina. 2024 Nov 1;44(11):1915-1922. doi: 10.1097/IAE.0000000000004201. PMID 39436300
- [Background] Szeto SKH, Lam JTW, Yu AHY, Pang CMK, Lin TPH, Hui VWK, Tsang KK, Chan JCK, Chen LJ, Lai TYY, Mohamed S, Tsang CW. Macular Hole Closure by Internal Limiting Membrane Flap without Gas Tamponade versus Conventional Surgery: A Comparative Study. Ophthalmol Retina. 2025 Nov;9(11):1034-1043. doi: 10.1016/j.oret.2025.06.005. Epub 2025 Jun 13. PMID 40518116
- [Background] Stopa M, Ciesielski M, Rakowicz P. Macular Hole Closure Without Endotamponade Application. Retina. 2023 Apr 1;43(4):688-691. doi: 10.1097/IAE.0000000000002850. Epub 2020 May 25. PMID 32453068